CLINICAL TRIAL: NCT07063446
Title: Integrating Corticospinal Tract Assessment Via sTMS And taVNS-Augmented CIMT In Infants With Hemiplegia
Brief Title: sTMS Combined With CIMT and taVNS In Infants With Hemiplegia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Dorothea Jenkins, Professor of Pediatrics, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00146198
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Hemiplegia; Perinatal Brain Injury
Keywords: constraint induced movement therapy; infants; taVNS; sTMS; hemiplegia
MeSH Terms: conditions — Hemiplegia

STUDY DESIGN:
Intervention Model Description: The trial is designed to use a diagnostic device prior to using an experimental treatment device paired with non-experimental physical therapy (CIMT).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- sTMS with taVNS paired CIMT (Experimental): sTMS diagnostic testing will be performed before and after 40hours of taVNS paired with CIMT treatment
  Interventions: Device: sTMS; Device: taVNS

INTERVENTIONS:
Device: sTMS — Single pulses of TMS will be delivered over the motor cortex to quantify and map the motor evoked potentials
Device: taVNS — taVNS will be used to stimulate the auricular branch of the vagus nerve and paired with CIMT for a total of 40hours of CIMT
  Other Names: transcutaneous auricular vagus nerve stimulation

SUMMARY:
Preterm and term infants with brain injury frequently have delayed motor skills, and one hand and arm may become stronger than the other, which can signal early cerebral palsy. A new treatment, transcutaneous vagus nerve stimulation (taVNS), boosts specific brain circuits and may improve function when paired with intensive motor activities. This study will test taVNS-paired constraint induced movement therapy in infants who have greater weakness on one side and determine if a single pulse of transcranial brain stimulation over the motor area can cause a measurable movement of the hand or thumb, and indicate which infants can benefit from 40h taVNS-paired CIMT.

DETAILED DESCRIPTION:
One of the most effective early therapies for improving motor skills in infants with unilateral motor weakness after perinatal brain injury, is constraint induced movement therapy (CIMT), in which a therapist engages a child in targeted play therapy with the more-affected arm/hand while the less-affected arm is immobilized in a mitt, reinforcing activity-dependent neuroplasticity. taVNS may accelerate functional gains and boost CIMT effects in young infants with hemiplegia over CIMT alone, based on pilot data. Before embarking on a larger scale trial, single pulse transcranial magnetic stimulation (sTMS) will be used to determine the connectivity and strength of the cortical spinal tract motor circuit with motor evoked potential of the hand or thumb.

The hypothesis is that the ability to respond to taVNS paired with intensive motor skill therapy in hemiplegic infants may be predicted by motor evoked potentials (MEP) elicited from sTMS over the motor cortex, as a quantifiable biomarker of CST circuit integrity, circuit response and cortical excitability.

ELIGIBILITY:
Inclusion Criteria:

* Infants 8-24mo with hemiplegia or asymmetric weakness of one arm, with or without truncal and transitional motor delays
* Gross Motor function Classification system (GMFCS) I - IV
* Parents are able to make consecutive appointments for assessments and intervention over 2wks and complete the 3mo follow-up.
* Parents are willing to fill out developmental questionnaires and provide the study team feedback on tolerability and outcomes.

Exclusion Criteria:

* previous CIMT within 3 months
* GMFCS V or severe motor impairment/quadriplegia
* uncorrected blindness/deafness, cardiomyopathy
* poorly controlled seizure disorder

Ages: 8 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Assisted Hand Assessment | 3months
  Percent Change in the mini-AHA or AHA from baseline to end of treatment- the standardized scale on the Assisted hand assessments range from 0-100 where 100 indicates greatest possible functional use of the hand and 0 indicates no hand function
Motor Evoked Potential (MEP) | 3 months
  Presence or absence (+ or -) of MEP in the affected upper extremity in response to sTMS of primary motor cortex in both hemispheres (circuit analysis)

SECONDARY OUTCOMES:
GMFM-88 | 3 months
  Percent Change in scores of Gross motor function measure-88 from baseline to end of treatment; total raw scores range from 0-264, with higher scores indicating greater motor function

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Videotapes of motor skills assessments are identifiable PHI and will not be shared. Extracted, de-identifed data may be shared on request.

REFERENCES:
- [Background] Sutter EN, Casey CP, Gillick BT. Single-pulse transcranial magnetic stimulation for assessment of motor development in infants with early brain injury. Expert Rev Med Devices. 2024 Mar;21(3):179-186. doi: 10.1080/17434440.2023.2299310. Epub 2024 Jan 3. PMID 38166497
- [Background] Casey CP, Sutter EN, Grimaldo A, Collins KM, Guerrero-Gonzalez J, McAdams RM, Dean DC 3rd, Gillick BT. Preservation of Bilateral Corticospinal Projections from Injured Hemisphere After Perinatal Stroke. Brain Sci. 2025 Jan 17;15(1):82. doi: 10.3390/brainsci15010082. PMID 39851449
- [Background] McGloon K, Humanitzki E, Brennan J, Summers P, Brennan A, George MS, Badran BW, Cribb AR, Jenkins D, Coker-Bolt P. Pairing taVNS and CIMT is feasible and may improve upper extremity function in infants. Front Pediatr. 2024 Feb 13;12:1365767. doi: 10.3389/fped.2024.1365767. eCollection 2024. PMID 38415207